CLINICAL TRIAL: NCT06590753
Title: Clinical and Radiographic Evaluation of the Effect of Osseodensefication Technique Versus Conventional Implant Drilling Technique on Supporting Structure in Implant Supported Mandibular Overdenture
Brief Title: Evaluation of the Effect of Osseodensefication Technique Versus Conventional Implant Drilling Technique in Implant Supported Mandibular Overdenture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Mai Ahmed Abdel Fatah, Dr., Badr University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1147620530
Record Dates: First submitted 2023-05-23; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Implant Site Reaction
Keywords: implant; Bone density; Bone height

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional (Active Comparator): One will be placed using the conventional drill method site preparation technique on one side of the mandible
  Interventions: Device: osseodensification bur
- osseodensification (Experimental): One will be placed using osseodensification (no cutting) implant site preparation technique on the other side.
  Interventions: Device: osseodensification bur

INTERVENTIONS:
Device: osseodensification bur — osseodensification bur

SUMMARY:
The present study will be performed to : evaluate the effect of two implant placement systems )conventional method and osseodensification method) radiographically on bone density and bone height surrounding the implant by using CBCT and clinically by probing depth and gingival index.

DETAILED DESCRIPTION:
Atrophic maxilla or mandible can lead to lack of prosthesis retention because of an inadequate bearing area causing both functional and physiological problems for patient, these problems can be treated for patient satisfaction with an implant supported fixed or removable complete or partial denture (1).

The use of implants to retain a mandibular over denture has been recommended as the first treatment choice for the edentulous mandible. From the available evidence; it shows that this treatment leads to a great improvement in both clinical function and patient's reported outcomes when compared to conventional complete dentures (2).

Clinical studies have reported that dental implants in the mandible have higher survival rates compared to those in the maxilla, having thinner cortical bone combined with thicker trabecular bone compared to the mandible (3). In contrast to the previous studies, additional studies in the posterior mandible showed high failure rates due to the poor bone quality as well as other additional factors (3-4).

The osseointegration process leads to new bone apposition on the implant surface and allows reaching the implant secondary stability that is the functional contact between living bone and titanium dental implant (4).

Primary implant stability is affected by both the quality and the quantity of bone of the osteotomy site. Hence, a precise evaluation of bone structure is essential before implant placement implant (5). The term bone quality depends on bone density, bone vascularity, bone metabolism and other factors that may affect implant outcome. Many authors describe bone density as being equivalent to bone quality. This includes physiological and structural parts and the degree of bone tissue mineralization (4-5).

2 Successful dental implant placement requires sufficient amount of bone thickness covering the implant so that primary stability is achieved, which is an important requirement for long term success of the implant (2, 6).

Primary implant stability is defined as the biomechanical stability upon implant insertion, being influenced by numerous factors, such as: bone quantity and quality, the geometric design of the implant, surgical technique, and insertion torque. From this stability, new bone develops around the surface of the implant, constituting a biological fixation named secondary implant stability (7, 8).

The longevity of any implant prosthesis depends on successful osseointegration and implant stability. Consistent osteotomies and densification are important to implant primary stability and to early loading (9, 10).

Unlike traditional bone drilling technologies, osseodensification does not excavate bone tissue. Rather, it preserves bone bulk, so bone tissue is simultaneously compacted and autografted in an outwardly expanding direction to form the osteotomy (11, 12). It creates a densified layer of surrounding bone through compaction autografting while simultaneously plastically expanding the bony ridge at the same time (13, 14,15).

The new burs allow bone preservation and condensation through compaction autografting during osteotomy preparation, increasing the peri-implant bone density (%BV), and the implant mechanical stability (16). .

Osseous densification was shown to increase the insertion and removal torques of the implants compared to standard drilling and extraction drilling. This demonstrates increased implant primary biomechanical stability (17).

3 Osseodensification had a direct impact on increasing the values of peak insertion torques of the implants compared to cutting drilling which indicates enhancement of initial stability of implant fixture (18).

ELIGIBILITY:
Inclusion Criteria:

* All patients will have edentulous.
* Patient's age ranges from 55-65 years.
* All patients should be free from any systemic disease such as bone diseases or debilitating diseases.
* Patient's residual ridge should be covered with firm mucosa free from any signs of inflammation, ulceration, or flabby tissue.
* Patients should have good oral hygiene.

Exclusion Criteria:

* Uncooperative patients will be excluded .
* Patient with parafunctional habits (bruxism, clenching)
* Patient with xerostomia or excessive salivation.
* Patient with TMJ disorder.

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
bone height | zero, 6, 12 months
  CBCT Measurements
bone density | zero, 6, 12 months
  CBCT Measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Azhar university (Grils), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No